CLINICAL TRIAL: NCT07067801
Title: Evaluation of Oral Corticosteroid Therapy in Idiopathic Sudden Unilateral Hearing Loss; a Randomized, Double Blind, Futility (Non-superiority) Trial.
Brief Title: Evaluation of Oral Corticosteroid Therapy in Idiopathic Sudden Unilateral Hearing Loss.
Acronym: ECOSUB
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Hôpital Civil de Strasbourg (Unknown); CHU de Reims (Other); Centre Hospitalo-Universitaire de Brabois, Vandoeuvre Les Nancy, France (Unknown); Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025/968
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Sudden Sensorineural Hearing Loss
Keywords: Sudden Sensorineural Hearing Loss; Corticosteroids; Randomized clinical trial; Placebo
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Fumigant 93

STUDY DESIGN:
Intervention Model Description: Randomized, controlled versus placebo, double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Placebo
- Oral Corticosteroid (Experimental): Standard of care
  Interventions: Drug: prednisone - oral corticosteroid 1mg/kg/D for 1 week

INTERVENTIONS:
Drug: prednisone - oral corticosteroid 1mg/kg/D for 1 week — Study of the Standard of care versus Placebo
  Arms: Oral Corticosteroid
Drug: Placebo — Control
  Arms: Control

SUMMARY:
Context: Idiopathic Sudden Sensorineural Hearing Loss (ISSHL) is a rapid-onset, sensorineural hearing loss of unknown etiology. It is one of the most common ENT emergencies, with spontaneous recovery occurring in 32% to 65% of cases. Treatment remains controversial, and the need for treatment itself is debated. Oral corticosteroids (OCS) are commonly used as first-line therapy, although they may have short-term side effects. Intratympanic corticosteroid injections (ITCIs) are an option for patients with contraindications to OCS or as a salvage treatment. The most recent Cochrane review includes three placebo-controlled studies on OCS efficacy (totaling 267 patients): two found no superiority of OCS, while one showed improvement in hearing. These studies are inconsistent and present methodological biases. Therefore, a sufficiently powered study is needed to assess OCS efficacy and establish clear treatment recommendations for ISSHL.

Objectives: Primary Objective: To demonstrate the equivalence of OCS as first-line treatment for ISSHL compared to no treatment, in terms of hearing recovery between days 7 and 10. Secondary Objectives: To assess the effect of OCS versus no treatment on tinnitus, and hearing recovery based on initial severity of ISSHL. To evaluate hearing recovery in patients treated with rescue ITCIs. In the absence of equivalence, to investigate the superiority of OCS over no treatment.

Methods: This multicenter, randomized, controlled equivalence trial will include two arms, each with 215 patients: one receiving OCS and the other a no-treatment control. In the absence of early hearing improvement, ITCIs will be administered regardless of study arm.

Perspective: The goal is to clarify the role of OCS in treating ISSHL and guide the development of updated treatment recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age
* ISSNH: idiopathic unilateral sensorineural hearing loss occurring in less than 72 hours, with loss of at least 30dB on 3 consecutive frequencies compared with the norm or the contralateral ear, confirmed on audiogram.
* Hearing loss beginning no more than 10 days ago
* Signed informed consent indicating that the subject has understood the purpose and procedures of the study, and agrees to participate in the study and to abide by its requirements and restrictions
* Affiliation with a French social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Otological medical history, illness or treatment affecting hearing
* Pregnancy
* Recurrent ISSNH
* Contraindication to oral corticosteroids or already treated with long-term corticosteroids
* Neurological symptoms other than vertigo or tinnitus
* Persons deprived of liberty by judicial or administrative decision; persons under forced psychiatric care; persons admitted to a health or social establishment for purposes other than research.
* Adults under legal protection or unable to express their consent
* Subjects who have been excluded from another study or who are on the "national volunteer list".
* Exclusion criteria during the course of the study : discovery of vestibular schwannoma, or other pathology explaining the SUB, on MRI centered on the internal auditory canals and cerebellopontine angles prescribed as part of routine care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Early hearing recovery | From enrollment to 10 +/- 2 days
  Hearing recovery defined by (composite criterion) :
  * Gain of at least 10dB in pure tone average (PTA) on pure tone audiometry compared with initial PTA in dB,
  * or > 10% improvement in intelligibility threshold on speech audiometry, compared with initial intelligibility threshold

SECONDARY OUTCOMES:
Medium-term hearing recovery | At 1 month and 3 months after enrollment
  Medium-term hearing recovery:
  * Gain of at least 10dB in pure tone average (PTA) on pure tone audiometry compared with initial PTA in dB,
  * or > 10% improvement in intelligibility threshold on speech audiometry, compared with initial intelligibility threshold
Tinnitus handicap | At 10 days, 1 month and 3 months after enrollment
  Change in tinnitus-related disability assessed by the Tinnitus Handicap Index (THI) score between inclusion and D10, M1, and M3.
Medium-term hearing recovery in patients without early recovery and treated with salvage trans-tympanic injections. | At 1 month and 3 months after enrollment
  Hearing recovery defined by (composite criterion) :
  * Gain of at least 10dB in pure tone average (PTA) on pure tone audiometry compared with initial PTA in dB
  * or > 10% improvement in intelligibility threshold on speech audiometry, compared with initial intelligibility threshold
Subgroup analysis based on initial severity | At 10 days, 1 month and 3 months after enrollment
  Subgroup analysis according to initial PTA ≥ 70dB or <70dB

CONTACTS AND LOCATIONS:
Overall Officials: Laurent TAVERNIER, MD PhD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be shared at the end of the study (> 3 years from now)
Access Criteria: IPD will be accessible upon request to the investigators of the study.